CLINICAL TRIAL: NCT01591421
Title: Phase I/II Study of the P13Kinase Inhibitor BKM120 Given in Combination With Panitumumab in Patients With Metastatic or Advanced RAS-Wild Type Colorectal Cancer.
Brief Title: P13Kinase Inhibitor BKM120 in Combination With Panitumumab in Metastatic/Advanced RAS-Wild Type Colorectal Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I208
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — NVP-BKM120; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BKM120 and Panitumumab (Experimental): BKM120 will be given either daily starting day 1 cycle 1or 5 out of 7 days every week, depending on when patient is enrolled on the study, in combination with panitumumab given intravenously every two weeks starting day 1 cycle 1.
  Interventions: Drug: BKM120; Drug: Panitumumab

INTERVENTIONS:
Drug: BKM120 — PO; Once daily starting day 1 cycle 1, or 5 out of 7 days every week.
Drug: Panitumumab — IV; Every two weeks starting day 1 cycle 1 (i.e. day 1 and 15 each 28 day cycle)

SUMMARY:
For the first phase of this study (phase I), the purpose will be to find the dose of a new drug, BKM120, that can safely be given in combination with standard dose panitumumab.

For the second phase of this study (phase II), the purpose is to find out what effects the combination of BKM120 and panitumumab, in doses found to be safe in the first part of the study, has on patients and their colorectal cancer.

DETAILED DESCRIPTION:
This is done by starting with doses of BKM120 at lower than the usual dose. Patients are given BKM120 and panitumumab and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then more patients are asked to join the study and are given higher doses of BKM120. If severe toxicity is seen, doses of BKM120 and/or panitumumab doses may be lowered in subsequent patients. Patients joining the study later on will normally get higher doses of BKM120 than patients who join earlier. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of a primary colorectal cancer which is recurrent or metastatic.
* Tumour must be confirmed to be K-Ras wild type (i.e. no K-Ras mutation found) by means of mutation analysis performed on representative samples of diagnostic tumour tissue by the standard regional or provincial laboratory and be eligible to receive standard panitumumab treatment as per local guidelines (i.e. must have failed, or have been unable to receive prior irinotecan, oxaliplatin and thymidylate synthase inhibitor therapy). Note: Archival tumour samples are acceptable for K-Ras mutation analysis.
* In the phase I portion of the trial, patients may have measurable OR non-measurable disease. Patients whose only evidence of disease progression is tumour marker elevation are not eligible.
* In the phase II portion of the trial, all patients must have measurable disease as defined by RECIST 1.1.

The criteria for defining measurable disease are as follows:

Chest X-ray ≥ 20 mm CT/MRI scan (with slice thickness of < 5 mm) ≥ 10 mm → longest diameter Physical exam (using calipers) ≥ 10 mm Lymph nodes by CT scan ≥ 15 mm → measured in short axis

Patients must have recovered from recent surgery, chemotherapy and/or radiation therapy and significant toxicity must have recovered to ≤ grade 2. At least 4 weeks must have elapsed from major surgery and radiation therapy, unless the radiation is low dose, does not involve mucosa and is non-myelosuppressive. Patient must have recovered (grade 0-1) from all reversible toxicity related to prior chemotherapy and have adequate washout from prior chemotherapy and investigational agents as follows: Washout period is the longest of one of the following:

1. two weeks
2. standard cycle length of prior regimen (i.e. 21 days for irinotecan q 3 weeks).
3. 10 half-lives for investigational drugs.

ECOG performance status of 0, 1 or 2.

* Laboratory Requirements: (must be done within 7 days prior to registration) Hematology: Absolute granulocytes (AGC) ≥ 1.0 x 109/L Platelets ≥ 100 x 109/L Hemoglobin ≥ 90 g/L Chemistry: Serum creatinine ≤ 1.5 x UNL OR Creatinine clearance ≥ 50 ml/min Bilirubin * ≤ UNL AST and ALT ≤ 3.0 x UNL Potassium ≤ UNL Calcium ≤ UNL Magnesium ≥ 0.5 mmol/L (may be achieved with supplementation) Blood glucose (fasting) < 7.8 mmol/L Coagulation: INR ≤ 2 x UNL (* direct, if patient known to have Gilberts)
* Patient must consent to provision of, and investigator(s) must confirm access to and agree to submit at the request of the NCIC CTG Central Tumour Bank, a representative formalin fixed paraffin block of tumour tissue in order that the correlative marker assays may be conducted. Where local centre regulations prohibit submission of blocks of tumour tissue, the approval of the NCIC CTG must be sought prior to registration of the first patient to allow a predetermined number of slides of representative tumour tissue to be substituted in response to the Central Tumour Bank request. Failure to submit any tissue samples on request will result in the patient being considered ineligible. Where no previously resected or biopsied tumour tissue exists, on the approval of the NCIC CTG, the patient may still be considered eligible for the study.
* Age ≥ 18 years. (Note that the lower age limit at each centre will be determined by that centre's policy regarding the age at which an individual may sign their own consent.)
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to registration. Patients of reproductive potential must agree to use highly effective contraception as follows:
* Female study subjects: during study and for 6 months after final dose of study therapy
* Male study subjects: during study and until 16 weeks after final dose of study therapy.
* Female partner of male study subject: during study and until 16 weeks after final dose of study therapy
* Patient consent for trial participation must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, standard consent forms for the trial will not be provided but sample forms are provided. A copy of the initial full board Research Ethics Board (REB) approval and approved consent forms must be sent to the central office. The patient must sign the consent forms prior to registration. Please note that the consent forms for this study must contain a statement which gives permission for qualified representatives of the CCTG, monitoring agencies and regulatory authorities to review patient records.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up. Patients enrolled in this trial must be treated and followed at the participating centre. This implies there must be a reasonable geographical limit (for example: 2 hour's driving distance) placed on the patients being considered for this trial.
* Protocol treatment is to begin within 5 working days of patient registration.

Exclusion Criteria:

* A history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 5 years.
* Women who are pregnant or breastfeeding.
* Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy (e.g. chronic pancreatitis, active chronic hepatitis, etc.).
* Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.
* Uncontrolled or significant cardiovascular disease including:

  * Myocardial infarction within 12 months;
  * Uncontrolled angina within 6 months;
  * Clinically significant congestive heart failure;
  * Stroke;
  * TIA or other ischemic event within 12 months;
  * Severe cardiac valve dysfunction
* Phase I: Patients may not be diabetic
* Phase II: Patients may be diabetic, but must have controlled diabetes (fasting glucose < 7.8 mmol/L)
* Patient has any of the following mood disorders:

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * ≥ CTCAE grade 3 anxiety
  * score of ≥ 10 in the PHQ-9
  * score of ≥ 15 in the GAD-7 mood scale
  * patient selects a positive response of '1, 2, 3' to question number 9 (suicidal ideation) in the PHQ-9
* Symptomatic metastases in the central nervous system. Subjects with signs or symptoms suggestive of brain metastasis are not eligible unless brain metastases are ruled out by CT or MRI scans.
* Patients who have received prior EGFR or PI3 Kinase inhibitor therapy.
* Receipt of an investigational therapeutic agent within washout period defined in section 5.1.4 of the protocol.
* Severe restrictive lung disease or radiological pulmonary findings of "interstitial lung disease" on the baseline chest x-ray which, in the opinion of the investigator, represents significant pathology.
* Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients who are unable to swallow capsules.
* Patients on potent CYP3A Inhibitors/Inducers (must have discontinued > 7 days prior to day 1) or therapeutic doses of warfarin like anticoagulants. Patients may receive low molecular weight heparin if indicated.
* Patients receiving chronic treatment with steroids or another immunosuppressive agent. Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients who are on a stable low dose corticosteroids treatment (e.g. dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible.
* Ongoing ocular inflammation or infection.
* Patients with significant (> grade 2) symptomatic ophthalmologic abnormalities such as:

  * Severe dry eye syndrome
  * Keratoconjunctivitis sicca
* Patients with known HIV (testing not mandatory) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of BKM120 (Phase I Component) | 24 months
  Determine the safety, tolerability, toxicity profile and dose limiting toxicities of BKM120 and Panitumumab.

SECONDARY OUTCOMES:
Anti-tumour activity (Phase II Component) | 24 months
  To assess the anti-tumour activity of BKM120 in combination with panitumumab as evidenced by response rates and early progression rates in patients with K-RAS wild-type metastatic colorectal cancer.
Translational Research | 24 months
  To investigate the correlation, if any, between response and molecular biomarkers in archival FFPE tumour.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, Study Chair — Ottawa Health Research Institute - General Division
Locations (3):
- Canada (3):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goodwin R, Jonker D, Chen E, Kennecke H, Cabanero M, Tsao MS, Vickers M, Bohemier C, Lim H, Ritter H, Tu D, Seymour L. A phase Ib study of a PI3Kinase inhibitor BKM120 in combination with panitumumab in patients with KRAS wild-type advanced colorectal cancer. Invest New Drugs. 2020 Aug;38(4):1077-1084. doi: 10.1007/s10637-019-00814-3. Epub 2019 Sep 10. PMID 31506897